CLINICAL TRIAL: NCT06687655
Title: Impact of Exogenous Ketones on Sleep Disruption in Vulnerable Populations: Phase 2 Study (KETO-SLEEP 2)
Brief Title: Impact of Exogenous Ketones on Sleep Apnea
Acronym: KETO-SLEEP 2
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: HVMN Inc (Industry); KETONE-IQ (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00439273-2
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea; Sleep
Keywords: sleep apnea; ketones; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Ketosis

STUDY DESIGN:
Intervention Model Description: The investigators will examine the preliminary efficacy of ingesting exogenous ketones before sleep on OSA. Patients with known OSA will be asked to temporarily discontinue CPAP, a technique used in our laboratory to temporarily elicit OSA. Prior to sleep the participants will ingest Ketone-IQ (20 g to 40 g - dose to be determined by KETO-SLEEP 1 trial), or placebo. Sleep will be assessed using a home sleep test (NOX T3) and questionnaires. Glucose will be monitored using a continuous glucose monitor (CGM).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone-IQ first (Experimental): This is a crossover study where participants will ingest either Ketone-IQ for 2 nights, or placebo for 2 nights before sleep. This arm will ingest Ketone-IQ first, then placebo.
  Interventions: Dietary Supplement: Ketone-IQ; Dietary Supplement: Placebo
- Placebo first (Experimental): This is a crossover study where participants will ingest either Ketone-IQ for 2 nights, or placebo for 2 nights before sleep. This arm will ingest Placebo first, then Ketone-IQ.
  Interventions: Dietary Supplement: Ketone-IQ; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone-IQ — This is a crossover study where participants will ingest either Ketone-IQ for 2 nights, or placebo for 2 nights before sleep. This is the Ketone-IQ (1,3 Butanediol) intervention.
Dietary Supplement: Placebo — This is a crossover study where participants will ingest either Ketone-IQ for 2 nights, or placebo for 2 nights before sleep. This is the Placebo intervention.

SUMMARY:
Obstructive Sleep Apnea (OSA) is a common medical disorder that is associated with reduced quality of life and higher risk of cardiovascular disease. Treatments for OSA and limited and not well tolerated. The investigator's lab has shown that a low carbohydrate, high fat ketogenic diet (KD) can reduce OSA severity. Since it can be challenging to adhere to a ketogenic diet, the investigators propose that ingesting exogenous ketones can be an alternative method to improve OSA. Specifically the investigators will examine the effect of taking a commercially available product (Ketone-IQ) at bedtime on overnight ketones and sleep quality. The investigators will also examine the effect of Ketone-IQ on sleep apnea severity, compared to placebo.

This project will examine the the preliminary efficacy of ingesting exogenous ketones before sleep on sleep apnea.

DETAILED DESCRIPTION:
Sleep is a vulnerable period during which blunted respiratory drive and low airway muscle tone can cause dangerous breathing disorders. Obstructive sleep apnea (OSA) describes the intermittent collapse of the upper airway that induces O2 desaturations and arousals from sleep, placing patients at risk for cardiovascular disease, stroke, and death. In some obese patients, sleep causes carbon dioxide (CO2) accumulation progressing to daytime hypercapnia, a condition called obesity hypoventilation syndrome (OHS). Continuous positive airway pressure (CPAP) treats OSA and OHS, but is poorly tolerated, and may not fully correct sleep dysfunction.

Changes in metabolism may help to control OSA or OHS. The investigators recently published results from the Ketogenic Diet for OHS clinical trial (KETOHS, NCT04108819) showing that a 2-week ketogenic diet (high fat, low carbohydrate) for patients with OSA and OHS lowered reduced CO2, serum bicarbonate (HCO3), respiratory quotient, nocturnal hypoxemia(2). KD also significantly improved OSA. After participants resumed prior diet, CO2 returned to baseline. The mechanisms by which KD improves sleep in this population could be related to reduced CO2 production (through fat oxidation), lowering of body weight, or direct effects of ketone bodies on sleep and breathing.

It is difficult to adhere long-term to KD, and there are multiple effects of this diet that make it challenging to understand mechanistic impacts on respiration. The investigators hypothesize that increasing ketone levels in the body, without having to adhere to a ketogenic diet, may be another method to improve breathing during sleep. Indeed, some drugs affecting acid-base status (e.g. acetazolamide or sulthiame) improve OSA, presumably through increasing and stabilizing respiratory drive. In this pilot study, the investigators will examine the pharmacokinetics, tolerability, and impacts of ingesting exogenous ketones (which are commercially available products) on sleep and breathing.

The specific ketone product to be tested for its impact on sleep and breathing is 1,3 butanediol (1,3BD) in a commercially available formulation called "Ketone IQ". 1,3BD is converted by liver metabolism into the ketone body beta-hydroxybutyrate (BHB) and has been utilized in multiple studies.

This project will be conducted in two studies, KETO-SLEEP 1 (KS1), and KETO-SLEEP 2 (KS2).

KETO-SLEEP 1: Examine the pharmacokinetics, tolerability, and sleep impacts of ingesting exogenous ketones (EK) before sleep (n=20, 10 men, 10 women). KS1 will lay the foundation for KS2 and other studies that administer exogenous ketones at bedtime, through dose-finding and assessment of tolerability. Patients with moderate-severe OSA (apnea-hypopnea index (AHI) >15)) adherent to CPAP will ingest EK or placebo 30 minutes before sleep. The participants will measure capillary BHB levels before ingestion and at 1, 3, 5, hours post-ingestion as well as upon awakening. CPAP use will be maintained on all nights and sleep architecture will be monitored with portable EEG. Questionnaires will solicit feedback about EK palatability, GI side effects, and sleep quality. Two doses (20 g and 40 g) of Ketone-IQ will be tested each for two nights, with one night used to measure BHB levels and separate night to allow for uninterrupted sleep.

KETO-SLEEP 2: Examine the preliminary efficacy of ingesting exogenous ketones before sleep on OSA (n=20, 10 men, 10 women). KS2 will examine the respiratory effects of exogenous ketones taken before sleep. Patients with known OSA will be asked to temporarily discontinue CPAP, a technique used in the investigator's laboratory to temporarily elicit OSA(10). To account for night-to-night variability in OSA severity the investigators will use portable sleep monitoring to collect sleep and respiratory data two nights under each condition. The dose of Ketone-IQ to be administered each night will vary from 20 to 40 g, depending upon results of KS-1.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-65 years old with a BMI of 18 - 35 kg/m2
2. History of moderate-severe OSA as defined by AHI >15 events/hr (American Academy of Sleep Medicine criteria),
3. Adherent to CPAP (objectively determined via device download over last 30 days) using CPAP at least 70% of days for >=4 hours.
4. CPAP pressure ≤10 cm water (H2O) (based on prescribed CPAP pressure, or median pressure on an auto-titrating CPAP device).

Exclusion Criteria:

1. No concomitant sleep disorder (such as insomnia, restless leg syndrome, narcolepsy, idiopathic hypersomnia)
2. No current daytime respiratory impairment such as uncontrolled asthma, or uncontrolled chronic obstructive pulmonary disease (COPD), pneumonia, interstitial lung disease.
3. No use of supplemental oxygen.
4. Currently on a low carbohydrate (<130 g carbohydrate/day) or ketogenic diet, intermittent fasting, or consuming exogenous ketones
5. Pregnancy or breastfeeding
6. Alcohol consumption of > 10 standard drinks per week
7. Use of nightly medications that affect breathing (e.g. opiates, acetazolamide)
8. Use of Sodium-glucose cotransporter-2 (SGLT2) inhibitors. For example, Canagliflozin (Invokana), Dapagliflozin (Farxiga), Empagliflozin (Jardiance), Ertugliflozin (Steglatro)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-09-06 (Estimated); Primary Completion 2028-09-06 (Estimated); Study Completion 2028-09-06 (Estimated)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI) | 2 nights Ketone-IQ, 2 nights Placebo
  Sleep studies will be performed using NOX T3 devices at home. The device will be worn for 2 consecutive nights during each intervention (Ketone IQ, Placebo); 4 nights total (2 nights Ketone-IQ, 2 nights Placebo). Apnea hypopnea index (AHI); mean number of apnoeas and hypopnoeas per hour of sleep will be calculated from NOX T3 data.

SECONDARY OUTCOMES:
Gastrointestinal Symptoms Questionnaire | 2 mornings after Ketone-IQ, 2 mornings after Placebo
  A questionnaire about gastro-intestinal symptoms will be administered each morning; 4 times total (2 mornings after Ketone-IQ, 2 mornings after Placebo). The instrument has 4 questions about upper GI symptoms, 4 questions about lower GI symptoms, and 4 questions about systemic symptoms. All questions are scored from 0 (no symptoms) to 8 (unbearable) for a score range of 0-96 (higher score = worse outcome).
Sleep-Related Impairment (SRI) as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS-SRI 8a) | 2 mornings after Ketone-IQ, 2 mornings after Placebo
  Sleep related impairment will be assessed by PROMIS-SRI 8a. Two mornings after Ketone-IQ, 2 mornings after Placebo; 4 nights total. A T-score is calculated from a raw score using conversion tables on the PROMIS website. The T-score (range 0-100) indicates the level of sleep-related impairment, with higher scores representing greater impairment
Sleep Disturbance (SD) as assessed by the PROMIS SD | 2 mornings after Ketone-IQ, 2 mornings after Placebo
  The PROMIS SD uses a 5-point Likert scale composed of eight items rated from 1 (not at all, very poor, or never) to 5 (very much, always, or very good) with four items reversed scored. Total raw scores range from 8 to 40 with higher scores indicating greater disturbance. Sleep disturbance will be measured a total of 4 times (2 mornings after Ketone-IQ, 2 mornings after Placebo)
Stanford Sleepiness Scale (SSS) | 2 mornings after Ketone-IQ, 2 mornings after Placebo
  The SSS consists of only one item. The scale requires respondents to select one of seven statements best representing their level of perceived sleepiness. Respondents use a scale from 1 to 7 to indicate their current level of sleepiness from 1 (feeling active and vital) - 7 (almost in reverie). Measured a total of 4 times (2 mornings after Ketone-IQ, 2 mornings after Placebo).
Oxygen Saturation Level | 2 nights on Ketone IQ, 2 nights on placebo
  NOX T3 data will be used to calculate metrics of oxygen saturation including mean oxygen level; measured a total of 4 times (2 nights on Ketone IQ, 2 nights on placebo).
Nadir Oxygen Level | 2 nights on Ketone IQ, 2 nights on placebo
  NOX T3 data will be used to calculate nadir oxygen level. Measured a total of 4 times (2 nights on Ketone IQ, 2 nights on placebo)
Oxygen Desaturation Index | 2 nights on Ketone IQ, 2 nights on placebo
  NOX T3 data will be used to calculate oxygen desaturation index. Measured a total of 4 times (2 nights on Ketone IQ, 2 nights on placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Jun, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Experimental data, including sleep data, questionnaires, and BHB measurements, will be stored as raw files on internal servers with cloud backup. Questionnaire data will be securely stored at Johns Hopkins University for three years post-study. Dr. Jun will control access to physical documents.
  Documentation and Accessibility: Research protocols, instrument details, and analysis methods will be detailed in publications. Deidentified data from published studies will be available at publication, accompanied by a data dictionary, and preserved for at least five years. Standard software (Excel, R, SPSS, SAS) will be used for data access and analysis.
Supporting Information: Study Protocol
Time Frame: Deidentified scientific data included in published manuscripts will be made available at the time of publication and additional data will be made available to researchers upon request. Data will be made available for up to 3 years following study completion.
Access Criteria: To request access to the data, researchers will be able to contact Dr. Jonathan Jun via email. Any data attached as a supplement to publications will be available for download from the publisher's website. The intention is to allow qualified external investigators broad access to the study data for specified research purposes.